CLINICAL TRIAL: NCT00522626
Title: Fetal Neurobehavior in Non-methadone Maintained Women in Substance Abuse Treatment
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lauren M. Jansson, Associate Professor of Pediatrics, Johns Hopkins University
Other Study IDs: 1490; R01DA019934 (NIH)
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy; Drug Abuse
Keywords: Fetus; Drug abuse; Fetal development; Substance abuse; Opioids; Methadone
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Opioid exposed pregnancies
  Interventions: Device: Maternal fetal monitoring

INTERVENTIONS:
Device: Maternal fetal monitoring — Simultaneous monitoring of maternal and fetal physiology
  Other Names: Toitu 325

SUMMARY:
This study seeks to elucidate fetal neurobehavioral development in fetuses of opioid dependent women who have either undergone and completed methadone detoxification,or who never received methadone maintenance, and are not methadone maintained at 36 weeks gestation. This research will determine how fetal neurobehavioral functioning in fetuses of opioid dependent, non-methadone maintained women differs from that of fetuses whose opioid dependent mothers are methadone maintained. The project will utilize a state-of-the-art computerized fetal actocardiograph and data analysis program to simultaneously evaluate fetal movement and heart rate, the interaction between the two and maternal physiologic parameters.

DETAILED DESCRIPTION:
This project examines fetal neurobehavior in non-methadone maintained, opioid dependent women. Subjects are outpatients at the Center for Addiction and Pregnancy on the Johns Hopkins Bayview Medical Center campus, who are between the ages of 18 and 40, who have either completed a methadone detoxification prior to 32 weeks gestation and are on no opiate replacement therapy after 32 weeks gestation, or who have never received methadone maintenance, and are free of maternal or known fetal health complications. Women are consented at 32 weeks of gestation. During the four weeks between consent and fetal testing, women will be privately interviewed by project staff and administered the SCLR-90 (Symptom Checklist) ASRS (Adult ADHD Self-Report Scale), and the PSD (Posttraumatic Stress Diagnostic Scale). These tools will be used to detect symptoms in different psychological domains (SCLR-90), ADHD (ASRS) and PTSD (PSD). At 36 weeks of gestation, women undergo fetal monitoring. Maternal demographic data (i.e. substance use history, pregnancy history, methadone dose, other medications) are abstracted from the maternal chart prior to each session. Women are asked a series of questions (the SOWS, or Subjective Opiate Withdrawal Scale and Adjective Questionnaire), via standardized questionnaires used to detect the presence or absence of withdrawal symptomatology prior to each session. Women will undergo two 60 minute fetal monitoring sessions on this day. The timing of the two sessions is such that it will provide two historical control groups. The first session will occur at 9 AM. The second session will occur at 1 P.M. The use of two fetal testing times will alleviate the problem of fetal circadian rhythms which would otherwise confound one or the other groups. The data acquisition is performed using a standard fetal monitoring system (Toitu 325). Data recorded include fetal movements and fetal heart rate. Additional data to be recorded include maternal EKG via 3 electrodes placed on the maternal chest (right mid sub-clavicle, left mid-axillary thorax) and upper left thigh (for ground lead), maternal respirations via a bellows apparatus attached around the maternal chest beneath the breasts, maternal contractions via the same transducer that detects fetal movement and fetal heart rate, and maternal skin conductance, or electrodermal activity via two electrodes with a gelled skin contact area placed on the index and middle fingers of one hand affixed with adhesive collars to limit gel contact to a 1 cm circle, and velcro. This maternal data will be time synchronized and analyzed in conjunction with fetal data. Also planned is the observation of fetal response to externally applied sound (a baby rattle). At the conclusion of the 60 minute session, an additional 6 minute recording will be added, with three sound stimuli at 1 minute intervals. Infants will undergo neurobehavioral testing on day #3 of life. This testing consists of the administration of the NICU Network Neurobehavioral Scale (the NNNS), a standardized 30-minute harmless and painless evaluation of the infant's motor, sensory and neurologic capabilities. The exam evaluates the infant's responses to auditory and visual stimuli, as well as movement, reflexes, signs of stress and consolability. Infants will also undergo an assessment for vagal tone on the first and third days of life. This assessment will involve obtaining 8-10 minutes of resting heart rate via 3 standard infant EKG leads while the infant is in a quiet state. The EKG leads will be connected directly to a Physio-control EKG monitor (R wave Medical Electronics of Florida). This reading is then transmitted to a vagal tone monitor (Delta Biometrics, Inc.) and computer for data storage and off-line analysis. Software will be used to computer heart period and vagal tone measures.

All fetal testing procedures obtained as part of this protocol are experimental; none are used for clinical purposes. Women consenting to participation will continue to receive routine care at CAP. Participants will be removed from the protocol if they should relapse to any licit or illicit substance between the time of consent (32 weeks gestation) and the time of fetal testing (36 weeks gestation).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women between ages 18 and 40, current clients of the CAP program
* Singleton, uncomplicated pregnancies, dated with routine 16 to 20 week ultrasound (as is part of standard care at CAP)
* Abstinence from licit and illicit substance abuse in the four weeks prior to consent

Exclusion Criteria:

* Complications of pregnancy, including gestational diabetes, polyhydramnios, hypertension, placenta previa or preterm labor
* Significant maternal health problems related to pregnancy, including HIV infection and Type I diabetes
* Significant maternal psychopathology or other pathology that would preclude informed consent (schizophrenia, mental retardation)
* Recent drug use, defined as positive urine toxicology (performed randomly at least weekly in the treatment center), clinical positives (subject appearing intoxicated at the treatment center) or patient report in the four weeks prior to recruitment, or at any time during study participation (i.e. from 28 weeks to 36 weeks gestation)
* Recent alcohol use, by clinical detection, patient report or breathalyzer reading (performed at the treatment center to confirm clinical impression) at any time in the four weeks prior to recruitment, or at any time during study participation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: OPioid exposed pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-08; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Jansson LM, Dipietro J, Elko A. Fetal response to maternal methadone administration. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):611-7. doi: 10.1016/j.ajog.2005.02.075. PMID 16150250
- [Result] Jansson LM, Di Pietro JA, Elko A, Williams EL, Milio L, Velez M. Pregnancies exposed to methadone, methadone and other illicit substances, and poly-drugs without methadone: a comparison of fetal neurobehaviors and infant outcomes. Drug Alcohol Depend. 2012 May 1;122(3):213-9. doi: 10.1016/j.drugalcdep.2011.10.003. Epub 2011 Oct 29. PMID 22041255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occured between May 2006 and May 2009 from a drug treatment facility treating pregnant and postpartum drug dependent women
Period: Overall Study
Arm/Group | Observational
Started | 19
Completed | 12
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Observational
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.25 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate
Description: Fetal heart rate in beats per minute
Time Frame: 60 minutes
Population: Total number of subjects completing assessment
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Trough Fetal Heart Rate: Opioid exposed pregnancies
Arm/Group | Trough Fetal Heart Rate
Number analyzed (Participants) | 12
beats per minute | 142.34 (10.60)

2. Secondary Outcome: Maternal Physiologic Parameters
Time Frame: 120 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Observational
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
Difficulty in recruiting leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No